CLINICAL TRIAL: NCT04390919
Title: Elevated Blood Monocyte Count Predicts 1 Year Poor Outcomes for Patients Admitted With Acute Decompensated Heart Failure
Brief Title: Prognostic Factors of Patients With ADHF
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, professor, Chongqing Medical University
Other Study IDs: 2020-05-04
Record Dates: First submitted 2020-05-04; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Acute Decompensated Heart Failure
Keywords: monocyte count; heart failure; acute decompensated heart failure; all-cause death
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high group: high group: monocyte count≥0.445×10*9 cells/L
  Interventions: Other: elevated monocyte count
- low group: low group: monocyte count<0.445×10*9 cells/L;

INTERVENTIONS:
Other: elevated monocyte count — The monocyte count at admission was higher than 0.445×10*9 cells/L
  Groups: high group

SUMMARY:
To explore the prognostic indicators for patients with ADHF

DETAILED DESCRIPTION:
According to ESC Guidelines for the diagnosis of acute heart failure 2008, patients with ADHF were diagnosed, and their medical history, laboratory examination and treatment plan were retrospectively analyzed, and the patients were followed up for 1 year. The 1-year outcomes of patients were analyzed to explore the prognostic indicators for patients with ADHF

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADHF diagnosed according to ESC Guidelines for the diagnosis of acute heart failure 2008

Exclusion Criteria:

* disorders of the hematopoietic system, history of cancer and/or previous treatment with chemotherapy, the infection caused by various pathogens, chronic inflammatory conditions, glucocorticoid therapy and/or histories of glucocorticoid use 3 months before the admission and acute myocardial infarction or coronary revascularization within the past 6 months. Also, patients who did not have a differential WBC count or who were lost to follow-up were excluded.

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ADHF patient diagnosed in the department of cardiovascular medicine in the first affiliated hospital of chongqing medical university
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2011-08-02 (Actual); Primary Completion 2015-02-16 (Actual); Study Completion 2015-02-16 (Actual)

PRIMARY OUTCOMES:
all-cause death | 1 year
  The primary end point was one-year all-cause death

SECONDARY OUTCOMES:
HF-related rehospitalization | 1 year
  the secondary end point was one-year HF-related rehospitalization.

IPD SHARING:
Plan to Share IPD: Undecided